CLINICAL TRIAL: NCT03640481
Title: A Phase 2, Randomized, Multicenter Study to Evaluate the Efficacy and Safety of KD025 in Subjects With Chronic Graft Versus Host Disease (cGVHD) After At Least 2 Prior Lines of Systemic Therapy (The ROCKstar Study)
Brief Title: Efficacy and Safety of KD025 in Subjects With cGVHD After At Least 2 Prior Lines of Systemic Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The sponsor has decided to prematurely terminate the study due to the challenges encountered in recruiting adolescent participants. This decision was made without any safety concerns.
Sponsor: Kadmon, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DRI17633; KD025-213 (Other: Kadmon); U1111-1279-2518 (Registry Identifier: ICTRP); DRI17633 (Other: Sanofi Identifier)
Record Dates: First submitted 2018-08-13; First posted 2018-08-21 (Actual); Results first posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-11

CONDITIONS: Chronic Graft-versus-host-disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — belumosudil; KD025

STUDY DESIGN:
Intervention Model Description: Phase 2, open label, randomized, multicenter study in subjects with cGVHD who have previously been treated with at least 2 prior lines of systemic therapy
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A: belumosudil 200 mg, QD, adult arm (Experimental): Eligible subjects randomized to arm A will take belumosudil 200 mg once daily
  Interventions: Drug: Belumosudil (KD025)
- Arm B: belumosudil 200 mg, BID, adult arm (Experimental): Eligible subjects randomized to arm B will take belumosudil 200 mg twice daily
  Interventions: Drug: Belumosudil (KD025)
- Adolescent arm A: belumosudil 200 mg QD (Experimental): Eligible subjects randomized to arm A will take belumosudil 200 mg once daily
  Interventions: Drug: Belumosudil (KD025)
- Adolescent arm B: belumosudil 200 mg BID (Experimental): Eligible subjects randomized to arm B will take belumosudil 200 mg twice daily
  Interventions: Drug: Belumosudil (KD025)

INTERVENTIONS:
Drug: Belumosudil (KD025) — Belumosudil is an orally available Rho-associated protein kinase-2 (ROCK2) selective inhibitor.
  Other Names: REZUROCK

SUMMARY:
This is a Phase 2, randomized, multicenter study to evaluate the efficacy and safety of KD025 in subjects with Chronic Graft Versus Host Disease (cGVHD) after at least 2 prior lines of systemic therapy

DETAILED DESCRIPTION:
Phase 2, open label, randomized, multicenter study in subjects with cGVHD who have previously been treated with at least 2 prior lines of systemic therapy. Approximately 166 subjects with active cGVHD will be randomized (1:1) to receive treatment with one of two belumosudil (formerly known as KD025) regimens:

* Arm A: belumosudil 200 mg QD
* Arm B: belumosudil 200 mg BID

With Amendment 2, the sample size was increased from approximately 126 subjects, with additional subjects to be enrolled as follows:

* 20 adolescents
* 20 adults into a site-specific Companion Study to collect biospecimens

These additional subjects will also be randomized (1:1) to Arm A or Arm B.

Any adolescent taking a proton pump inhibitor (PPI) or a strong CYP3A4 inducer will begin Cycle 1 Day 1 at the escalated dose of belumosudil 200 mg BID.

Randomization will be stratified according to prior cGVHD treatment with ibrutinib (Yes / No) and severe cGVHD at baseline (Yes / No). Subjects may receive treatment in 28-day treatment cycles until clinically significant progression of cGVHD. Subjects who have not achieved a response after 12 cycles of belumosudil should be withdrawn if in the Investigator's judgment there is no evidence of clinical benefit. Subjects will undergo evaluations as outlined in the Study Assessments table (Appendix A). The primary endpoint is the overall response rate (ORR) with responses as defined by the 2014 National Institute of Health (NIH) Consensus Development Project on clinical trials in cGVHD.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects at least 12 years of age who have had allogenic hematopoietic cell transplant (HCT).
2. Previously received at least 2 and not more than 5 lines of systemic therapy for cGVHD
3. Receiving glucocorticoid therapy with a stable dose over the 2 weeks prior to screening
4. Have persistent cGVHD manifestations and systemic therapy is indicated
5. Karnofsky Performance Score of ≥ 60 (if aged 16 years or older); Lansky Performance Score of ≥ 60 (if aged < 16 years)
6. Weight ≥ 40kg

Exclusion Criteria:

1. Subjects has not been on a stable dose / regimen of systemic cGVHD treatments for at least 2 weeks prior to screening. (Note: Concomitant corticosteroids, calcineurin inhibitors, sirolimus, MMF, methotrexate, rituximab, and extracorporeal photophoresis (ECP) are acceptable. Systemic investigational GVHD treatments are not permitted).
2. Histological relapse of the underlying cancer or post-transplant lymphoproliferative disease at the time of screening.
3. Current treatment with ibrutinib. Prior treatment with ibrutinib is allowed with a washout of at least 28 days prior to randomization.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (35):
- United States (35):
  - Phoenix Childrens Hospital Site Number : 154, Phoenix, Arizona
  - University of Arizona - Cancer Center Site Number : 122, Tucson, Arizona
  - City of Hope Medical Center Site Number : 050, Duarte, California
  - University of California, Los Angeles (UCLA) - Medical Center Site Number : 104, Los Angeles, California
  - University of California, San Francisco (UCSF) - Helen Diller Family Comprehensive Cancer Center Site Number : 058, San Francisco, California
  - Stanford Cancer Center Site Number : 108, Stanford, California
  - Colorado Blood Cancer Institute Site Number : 098, Denver, Colorado
  - University of Miami - Sylvester Cancer Center Site Number : 097, Miami, Florida
  - Moffitt Site Number : 102, Tampa, Florida
  - Emory University School of Medicine Site Number : 100, Atlanta, Georgia
  - Augusta University Medical Center Site Number : 093, Augusta, Georgia
  - University of Illinois at Chicago Site Number : 139, Chicago, Illinois
  - University of Iowa Site Number : 126, Iowa City, Iowa
  - University of Kansas Cancer Center Site Number : 105, Fairway, Kansas
  - Center for Cancer Research National Cancer Institute Site Number : 107, Bethesda, Maryland
  - Massachusetts General Hospital Site Number : 002, Boston, Massachusetts
  - Dana-Farber Cancer Institute Site Number : 004, Boston, Massachusetts
  - CS Mott Children's Hospital Site Number : 157, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute-4100 John R St Site Number : 094, Detroit, Michigan
  - University of Minnesota Site Number : 051, Minneapolis, Minnesota
  - Washington University School of Medicine Site Number : 125, St Louis, Missouri
  - University of Rochester Site Number : 106, Rochester, New York
  - Wake Forest Site Number : 123, Winston-Salem, North Carolina
  - The Cleveland Clinic Foundation Site Number : 041, Cleveland, Ohio
  - James Cancer Hospital & Wexner Medical Center at the Ohio State University Comprehensive Cancer Center Site Number : 103, Columbus, Ohio
  - Oregon Health & Science University (OHSU) Site Number : 095, Portland, Oregon
  - University of Pittsburgh Medical Center (UPMC) - Hillman Cancer Center Site Number : 132, Pittsburgh, Pennsylvania
  - Sarah Cannon and HCA Research Institute Site Number : 007, Nashville, Tennessee
  - Vanderbilt University Medical Center Site Number : 063, Nashville, Tennessee
  - South Austin Medical Center Site Number : 091, Austin, Texas
  - MD Anderson Cancer Center Site Number : 057, Houston, Texas
  - Texas Transplant Institute Site Number : 079, San Antonio, Texas
  - Fred Hutchinson Cancer Research Center Site Number : 052, Seattle, Washington
  - University of Wisconsin - Carbone Cancer Center Site Number : 135, Madison, Wisconsin
  - Froedtert Hospital and the Medical College of Wisconsin Site Number : 101, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org.

REFERENCES:
- [Background] Przepiorka D, Le RQ, Ionan A, Li RJ, Wang YH, Gudi R, Mitra S, Vallejo J, Okusanya OO, Ma L, Yang Y, Patel P, Mezaache D, Shah R, Banerjee A, McLamore S, Maung AN, Goldberg KB, Pazdur R, Theoret MR, De Claro RA. FDA Approval Summary: Belumosudil for Adult and Pediatric Patients 12 Years and Older with Chronic GvHD after Two or More Prior Lines of Systemic Therapy. Clin Cancer Res. 2022 Jun 13;28(12):2488-2492. doi: 10.1158/1078-0432.CCR-21-4176. PMID 35135839
- [Derived] Sharma R, Holtzman NG, Pusic I, Cutler C, Treister N, Mehta RS, Alousi AS, Vigneswaran N, Javaid A, Boksa F, Mody DP, Costa-da-Silva AC, Schueller O, Mace S, Yao Y, Ji R, Hu B, Marshall K, Blazar BR, Lee SJ, Pavletic SZ, Mays JW. Belumosudil reduces oral chronic graft-versus-host disease tissue inflammation and fibrosis: a ROCKstar companion study. Blood Adv. 2025 Jul 22;9(14):3479-3494. doi: 10.1182/bloodadvances.2025016170. PMID 40311075
- [Derived] Lee SJ, Cutler C, Blazar BR, Tu A, Yang Z, Pavletic SZ. Correlation of Patient-Reported Outcomes with Clinical Organ Responses: Data from the Belumosudil Chronic Graft-versus-Host Disease Studies. Transplant Cell Ther. 2022 Oct;28(10):700.e1-700.e6. doi: 10.1016/j.jtct.2022.06.020. Epub 2022 Jul 1. PMID 35781099
- [Derived] Cutler C, Lee SJ, Arai S, Rotta M, Zoghi B, Lazaryan A, Ramakrishnan A, DeFilipp Z, Salhotra A, Chai-Ho W, Mehta R, Wang T, Arora M, Pusic I, Saad A, Shah NN, Abhyankar S, Bachier C, Galvin J, Im A, Langston A, Liesveld J, Juckett M, Logan A, Schachter L, Alavi A, Howard D, Waksal HW, Ryan J, Eiznhamer D, Aggarwal SK, Ieyoub J, Schueller O, Green L, Yang Z, Krenz H, Jagasia M, Blazar BR, Pavletic S. Belumosudil for chronic graft-versus-host disease after 2 or more prior lines of therapy: the ROCKstar Study. Blood. 2021 Dec 2;138(22):2278-2289. doi: 10.1182/blood.2021012021. Erratum In: Blood. 2022 Mar 17;139(11):1772. doi: 10.1182/blood.2022015598. PMID 34265047

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 33 centers in the United States. A total of 251 participants were screened between 11 October 2018 to 08 August 2023, of which 92 participants were screen failures in adult cohort due to not meeting eligibility criteria, there were no screen failures in adolescent cohort.
Pre-assignment Details: 156 participants were randomized in the adult cohort, 4 of which did not receive treatment. 3 participants were randomized in the adolescent cohort. The sponsor decided to prematurely terminate the study due to the challenges encountered in recruiting adolescent participants. This decision was made without any safety concerns.
Groups:
- Adult Arm A: Belumosudil 200 mg QD: Participants received belumosudil 200 milligram (mg) tablet orally once a day (QD) in 28-day cycles until clinically significant progression of chronic graft versus host disease (cGVHD), histologic recurrence of underlying malignancy, unacceptable toxicity, Investigator decision, participant preference/withdrawal of consent, loss of follow-up, sponsor decision, or death (whichever occurred first).
- Adult Arm B: Belumosudil 200 mg BID: Participants belumosudil 200 mg tablet orally twice a day (BID) in 28-day cycles until clinically significant progression of cGVHD, histologic recurrence of underlying malignancy, unacceptable toxicity, Investigator decision, participant preference/withdrawal of consent, loss of follow-up, sponsor decision, or death (whichever occurred first).
- Adolescent Arm A: Belumosudil 200 mg QD: Participants received belumosudil 200 mg tablet orally QD in 28-day cycles until clinically significant progression of cGVHD, histologic recurrence of underlying malignancy, unacceptable toxicity, Investigator decision, participant preference/withdrawal of consent, loss of follow-up, sponsor decision, or death (whichever occurred first).
- Adolescent Arm B: Belumosudil 200 mg BID: Participants received belumosudil 200 mg tablet orally BID in 28-day cycles until clinically significant progression of cGVHD, histologic recurrence of underlying malignancy, unacceptable toxicity, Investigator decision, participant preference/withdrawal of consent, loss of follow-up, sponsor decision, or death (whichever occurred first).
Period: Overall Study
Arm/Group | Adult Arm A: Belumosudil 200 mg QD | Adult Arm B: Belumosudil 200 mg BID | Adolescent Arm A: Belumosudil 200 mg QD | Adolescent Arm B: Belumosudil 200 mg BID
Started | 78 | 78 | 2 | 1
Completed | 0 | 0 | 0 | 0
Not Completed | 78 | 78 | 2 | 1
Not completed — Death | 14 | 14 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0
Not completed — Site terminated by sponsor | 1 | 3 | 0 | 0
Not completed — Study terminated by sponsor | 29 | 42 | 1 | 0
Not completed — Withdrawal by Subject | 5 | 4 | 0 | 1
Not completed — Other | 26 | 12 | 1 | 0
Not completed — Randomized, but not treated | 1 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat (mITT) population included all randomized participants who received at least one dose of study drug.
Groups:
- Adult Arm A: Belumosudil 200 mg QD; Adolescent Arm A: Belumosudil 200 mg QD: Participants received belumosudil 200 mg tablet orally QD in 28-day cycles until clinically significant progression of cGVHD, histologic recurrence of underlying malignancy, unacceptable toxicity, Investigator decision, participant preference/withdrawal of consent, loss of follow-up, sponsor decision, or death (whichever occurred first).
- Adult Arm B: Belumosudil 200 mg BID: Participants belumosudil 200 mg tablet orally BID in 28-day cycles until clinically significant progression of cGVHD, histologic recurrence of underlying malignancy, unacceptable toxicity, Investigator decision, participant preference/withdrawal of consent, loss of follow-up, sponsor decision, or death (whichever occurred first).
- Total: Total of all reporting groups
Arm/Group | Adult Arm A: Belumosudil 200 mg QD | Adult Arm B: Belumosudil 200 mg BID | Adolescent Arm A: Belumosudil 200 mg QD | Adolescent Arm B: Belumosudil 200 mg BID | Total
Number analyzed (Participants) | 77 | 75 | 2 | 1 | 155
Age, Customized [Count of Participants; unit: Participants]
  12-17 Years | 0 | 0 | 2 | 1 | 3
  18-77 Years | 77 | 75 | 0 | 0 | 152
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 38 | 0 | 1 | 67
  Male | 49 | 37 | 2 | 0 | 88
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 0 | 0 | 2
  Asian | 2 | 2 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 1 | 1 | 0 | 9
  White | 65 | 67 | 1 | 1 | 134
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 0 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: The ORR was defined as the percentage of participants with a best response meeting the overall response criteria assessment of complete response (CR) or partial response (PR) at any post-baseline response assessment. CR was defined as resolution of all manifestations of cGVHD in each organ or site. PR was defined as the improvement in at least one organ or site without progression in any other organ or site. Responses were assessed by the 2014 National Institutes of Health (NIH) Consensus Development Project on Clinical Trials in cGVHD.
Time Frame: From the date of randomization to the date of first documentation of progression or death due to any cause or data cut-off, whichever occurred first (maximum duration: up to 40.5 months for adult arms and 27.6 months for adolescent arms)
Population: mITT population included all randomized participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Adult Arm A: Belumosudil 200 mg QD | Adult Arm B: Belumosudil 200 mg BID | Adolescent Arm A: Belumosudil 200 mg QD | Adolescent Arm B: Belumosudil 200 mg BID
Number analyzed (Participants) | 77 | 75 | 2 | 1
Percentage of participants | 74.0 | 76.0 | 50.0 | 100.0

2. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time from first documentation of response to the time of first documentation of deterioration from best response (e.g., CR to PR, or PR to Lack of response [LR]). CR was defined as resolution of all manifestations of cGVHD in each organ or site. PR was defined as the improvement in at least one organ or site without progression in any other organ or site. LR included the response status of mixed, unchanged, or progression. Mixed LR was defined as complete or partial response in at least one organ accompanied by progression in another organ. Unchanged LR was defined as outcomes that did not meet the criteria for complete response, partial response, progression or mixed response. Progression LR-P was defined as progression in at least one organ or site without a response in any other organ or site. Confidence interval (CI) is calculated using Kaplan-Meier method.
Time Frame: as for outcome 1
Population: Responder population included participants in the mITT population that achieved a partial or complete response at any post-baseline response assessment.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Adult Arm A: Belumosudil 200 mg QD | Adult Arm B: Belumosudil 200 mg BID | Adolescent Arm A: Belumosudil 200 mg QD | Adolescent Arm B: Belumosudil 200 mg BID
Number analyzed (Participants) | 57 | 57 | 1 | 1
Weeks | 23.9 [11.43 to 50.43] | 32.0 [20.86 to 53.14] | 16.1 [NA to NA] — NA indicates that confidence interval (CI) was not estimable due to insufficient number of participants with events at study closure. | 4.1 [NA to NA] — NA indicates that CI was not estimable due to insufficient number of participants with events at study closure.

3. Secondary Outcome: Number of Participants With Improvement (>=7-Point Reduction [7-PtR] From Baseline) as Assessed by Lee Symptom Scale (LSS) Score
Description: The questionnaire asked participants to indicate the degree of bother that they experienced due to symptoms in 7 domains potentially affected by chronic GVHD. It consists of 30 items of 7 domains: skin, eyes and mouth, breathing, eating and digestion, muscles and joints, energy, and mental and emotional. Each question is scored 0, 1, 2, 3 or 4. A domain score was calculated for each domain by taking the mean of all items completed if more than 50% were answered and normalizing to a 0 to 100 scale. A summary score was calculated as average of all non-missing domain scores if more than 50% of them were non-missing. A higher score indicated more bothersome symptoms. A 7-point difference on the summary score of cGVHD symptom scale was found to be clinically meaningful.
Time Frame: Baseline (Day 1) up to 40.5 months for adult arms; Baseline (Day 1) up to 27.6 months for adolescent arms
Population: mITT population included all randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Adult Arm A: Belumosudil 200 mg QD | Adult Arm B: Belumosudil 200 mg BID | Adolescent Arm A: Belumosudil 200 mg QD | Adolescent Arm B: Belumosudil 200 mg BID
Number analyzed (Participants) | 77 | 75 | 2 | 1
Participants | 45 | 48 | 0 | 0

4. Secondary Outcome: Number of Participants With Best Response by Organ System
Description: The best response (CR, PR) for individual organs (skin, eyes, mouth, esophagus, upper gastrointestinal [GI], lower GI, liver, lungs, joints and fascia) were summarized. CR was defined as resolution of all manifestations of cGVHD in each organ or site. PR was defined as the improvement in at least one organ or site without progression in any other organ or site.
Time Frame: From date of randomization until disease progression or data cut-off, whichever occurred first (maximum duration: up to 40.5 months for adult arms and 27.6 months for adolescent arms)
Population: mITT population included all randomized participants who received at least one dose of study drug. Only those participants with data collected for each specified category are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Adult Arm A: Belumosudil 200 mg QD | Adult Arm B: Belumosudil 200 mg BID | Adolescent Arm A: Belumosudil 200 mg QD | Adolescent Arm B: Belumosudil 200 mg BID
Number analyzed (Participants) | 63 | 63 | 2 | 1
Participants
  Skin: number analyzed (Participants) | 63 | 63 | 1 | 0
  Skin | 20 | 28 | 1 |
  Eyes: number analyzed (Participants) | 56 | 52 | 0 | 1
  Eyes | 24 | 26 |  | 1
  Mouth: number analyzed (Participants) | 41 | 51 | 1 | 1
  Mouth | 23 | 31 | 1 | 1
  Esophagus: number analyzed (Participants) | 23 | 13 | 0 | 0
  Esophagus | 13 | 7 |  |
  Upper GI: number analyzed (Participants) | 14 | 10 | 0 | 0
  Upper GI | 9 | 4 |  |
  Lower GI: number analyzed (Participants) | 7 | 8 | 0 | 0
  Lower GI | 5 | 6 |  |
  Liver: number analyzed (Participants) | 10 | 4 | 0 | 0
  Liver | 2 | 1 |  |
  Lungs: number analyzed (Participants) | 27 | 25 | 2 | 0
  Lungs | 9 | 6 | 0 |
  Joints and Fascia: number analyzed (Participants) | 59 | 57 | 0 | 0
  Joints and Fascia | 42 | 39 |  |

5. Secondary Outcome: Percentage of Participants With Best Response of PR and CR
Description: PR was defined as the improvement in at least one organ or site without progression in any other organ or site. CR was defined as resolution of all manifestations of cGVHD in each organ or site. Responses were assessed by the 2014 NIH Consensus Development Project on Clinical Trials in cGVHD.
Time Frame: as for outcome 1
Population: mITT population included all randomized participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Adult Arm A: Belumosudil 200 mg QD | Adult Arm B: Belumosudil 200 mg BID | Adolescent Arm A: Belumosudil 200 mg QD | Adolescent Arm B: Belumosudil 200 mg BID
Number analyzed (Participants) | 77 | 75 | 2 | 1
Percentage of participants
  PR | 68.8 | 73.3 | 50.0 | 100.0
  CR | 5.2 | 2.7 | 0 | 0

6. Secondary Outcome: Percent Change From Baseline in Corticosteroid Dose to Greatest Reduction
Description: Change in corticosteroid doses was analyzed by using prednisone dose equivalents. If participants were not using prednisone as the systemic corticosteroid, then the prednisone dose equivalent would be determined according to following conversion ratios: 1 mg prednisone is equivalent to: 4.0 mg Hydrocortisone; 0.8 mg Methylprednisolone; 0.15 mg Dexamethasone; 1.0 mg Prednisolone and 0.8 mg Triamcinolone.
Time Frame: Baseline (Day 1) and 40.5 months for adult arms; Baseline (Day 1) and 27.6 months for adolescent arms
Population: mITT population included all randomized participants who received at least one dose of study drug. Only those participants with data collected at specified timepoints are reported.
Measure: Median (Full Range); unit: Percent change
Arm/Group | Adult Arm A: Belumosudil 200 mg QD | Adult Arm B: Belumosudil 200 mg BID | Adolescent Arm A: Belumosudil 200 mg QD | Adolescent Arm B: Belumosudil 200 mg BID
Number analyzed (Participants) | 73 | 73 | 2 | 1
Percent change | -50.00 [-100.0 to 0.0] | -66.67 [-100.0 to 900.0] | -50.00 [-100.0 to 0.0] | -60.00 [-60.0 to -60.0]

7. Secondary Outcome: Percentage of Participants With Reduction and Discontinuation of Calcineurin Inhibitor Dose
Description: Calcineurin inhibitors include systemic tacrolimus and cyclosporine. Percentage of participants with reduction and discontinuation of calcineurin inhibitor dose is presented.
Time Frame: Baseline (Day 1) up to 40.5 months for adult arms; Baseline (Day 1) up to 27.6 months for adolescent arms
Population: mITT population included all randomized participants who received at least one dose of study drug. Only those participants who received CNI at baseline were included in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Adult Arm A: Belumosudil 200 mg QD | Adult Arm B: Belumosudil 200 mg BID | Adolescent Arm A: Belumosudil 200 mg QD | Adolescent Arm B: Belumosudil 200 mg BID
Number analyzed (Participants) | 32 | 26 | 1 | 0
Percentage of participants
  Reduction of Calcineurin Inhibitor Dose | 46.9 | 57.7 | 100.0 |
  Discontinuation of Calcineurin Inhibitor Dose | 21.9 | 34.6 | 0 |

8. Secondary Outcome: Failure-Free Survival (FFS)
Description: FFS was defined as the absence of new cGVHD systemic therapy, non-relapse mortality and recurrent malignancy (i.e. underlying disease) and was censored by last response assessment or long term follow up assessment, whichever was the latest and available.
Time Frame: From first dose of study drug to the time of first documentation of response or data cut-off, whichever occurred first (maximum duration: up to 40.5 months for adult arms and 27.6 months for adolescent arms)
Population: mITT population included all randomized participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Adult Arm A: Belumosudil 200 mg QD | Adult Arm B: Belumosudil 200 mg BID | Adolescent Arm A: Belumosudil 200 mg QD | Adolescent Arm B: Belumosudil 200 mg BID
Number analyzed (Participants) | 77 | 75 | 2 | 1
Months | 16.3 [10.15 to 26.48] | 17.2 [11.27 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of participants with events at study closure. | NA [NA to NA] — NA indicates that median and CI was not estimable due to insufficient number of participants with events at study closure. | 6.8 [NA to NA] — NA indicates that CI was not estimable due to insufficient number of participants with events at study closure.

9. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as time from first dose of belumosudil to the date of death due to any cause.
Time Frame: From first dose of study drug to date of death from any cause or data cut-off, whichever occurred first (maximum duration: up to 40.5 months for adult arms and 27.6 months for adolescent arms)
Population: mITT population included all randomized participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Adult Arm A: Belumosudil 200 mg QD | Adult Arm B: Belumosudil 200 mg BID | Adolescent Arm A: Belumosudil 200 mg QD | Adolescent Arm B: Belumosudil 200 mg BID
Number analyzed (Participants) | 77 | 75 | 2 | 1
Months | NA [NA to NA] — NA indicates that median and 95% CI was not estimable due to insufficient number of participants with events at study closure. | NA [NA to NA] — NA indicates that median and 95% CI was not estimable due to insufficient number of participants with events at study closure. | NA [NA to NA] — NA indicates that median and 95% CI was not estimable due to insufficient number of participants with events at study closure. | NA [NA to NA] — NA indicates that median and 95% CI was not estimable due to insufficient number of participants with events at study closure.

10. Secondary Outcome: Number of Participants With Best Response of Global Severity Rating Score as Based on the Clinician-Reported Global cGVHD Activity Assessment
Description: The Clinician-reported global cGVHD Activity Assessment is a 0-10 point numeric rating scale with a score of 0 indicating "cGVHD symptoms not at all severe" and a score of 10 being "most severe cGVHD symptoms possible". Higher scores indicated worse symptoms. Best response was defined as PR+CR. PR was defined as the improvement in at least one organ or site without progression in any other organ or site. CR was defined as resolution of all manifestations of cGVHD in each organ or site. Participants were categorized in 3 categories at baseline based on the global severity scores of <6, =6-7 and >7 and number of participants with best response for them is reported.
Time Frame: Baseline (Day 1) up to 40.5 months for adult arms; Baseline (Day 1) up to 27.6 months for adolescent arms
Population: mITT population included all randomized participants who received at least one dose of study drug. Only participants with respective global severity rating score categories of <6, =6-7 and >7 assessed at baseline are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Adult Arm A: Belumosudil 200 mg QD | Adult Arm B: Belumosudil 200 mg BID | Adolescent Arm A: Belumosudil 200 mg QD | Adolescent Arm B: Belumosudil 200 mg BID
Number analyzed (Participants) | 77 | 75 | 2 | 1
Participants
  Baseline global severity rating score < 6: Best response: number analyzed (Participants) | 22 | 16 | 1 | 1
  Baseline global severity rating score < 6: Best response | 9 | 8 | 0 | 0
  Baseline global severity rating score= 6-7: Best response: number analyzed (Participants) | 30 | 40 | 1 | 0
  Baseline global severity rating score= 6-7: Best response | 15 | 28 | 1 |
  Baseline global severity rating score >7: Best response: number analyzed (Participants) | 25 | 19 | 0 | 0
  Baseline global severity rating score >7: Best response | 11 | 9 |  |

11. Secondary Outcome: Change From Baseline in Patient Self-Reported Symptom Activity Based on cGVHD Activity Assessment
Description: The symptom activity item is a 0-10-point numeric rating scale with a score of 0 indicating "cGVHD symptoms not at all severe" and a score of 10 being "most severe cGVHD symptoms possible". The status reported by participants were categorized as none, mild, moderate, and severe. Higher scores indicated worse symptoms. Baseline was defined as the valid and last non-missing value obtained within 14 days prior to participants receiving the first study drug.
Time Frame: Baseline (Day 1) and 40.5 months for adult arms; Baseline (Day 1) and 27.6 months for adolescent arms
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Adult Arm A: Belumosudil 200 mg QD | Adult Arm B: Belumosudil 200 mg BID | Adolescent Arm A: Belumosudil 200 mg QD | Adolescent Arm B: Belumosudil 200 mg BID
Number analyzed (Participants) | 52 | 48 | 2 | 1
Score on a scale | -0.9 (2.4) | -1.5 (2.4) | 0.0 (0.0) | -1.0 (NA) — NA indicates that standard deviation could not be determined when only 1 participant was analyzed.

12. Secondary Outcome: Maximum Concentration Observed (Cmax) of Belumosudil
Description: Blood samples were collected at the specified timepoints to evaluate Cmax of belumosudil. As pre-specified in protocol, pharmacokinetic (PK) parameters were only calculated for participants with full PK samples. Thus, PK parameters were not calculated for adolescent participants who only had sparse PK samples.
Time Frame: Cycles 1 and 2: Pre-dose and 1, 2, 3, 4, 5, 6, 7, 8, and 12 hours post dose on Day 1 for adult arms; Cycles 2 and 4: Pre-dose and 3 and 5 hours post dose on Day 1 for adolescent arms
Population: PK population included all study participants who provided samples for dense PK sampling. Only those participants with data collected at specified timepoints are reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Adult Arm A: Belumosudil 200 mg QD | Adult Arm B: Belumosudil 200 mg BID | Adolescent Arm A: Belumosudil 200 mg QD | Adolescent Arm B: Belumosudil 200 mg BID
Number analyzed (Participants) | 5 | 5 | 2 | 1
Nanograms per milliliter (ng/mL)
  Cycle 1: number analyzed (Participants) | 5 | 5 | 0 | 0
  Cycle 1 | 1350 (127) | 870 (177) |  |
  Cycle 2: number analyzed (Participants) | 4 | 4 | 2 | 1
  Cycle 2 | 1780 (154) | 2050 (99.9) | NA (NA) — As pre-specified in protocol, Cmax was only calculated for participants with full PK samples. Thus, Cmax was not calculated for adolescent participants who only had sparse PK samples. | NA (NA) — As pre-specified in protocol, Cmax was only calculated for participants with full PK samples. Thus, Cmax was not calculated for adolescent participants who only had sparse PK samples.
  Cycle 4: number analyzed (Participants) | 0 | 0 | 2 | 1
  Cycle 4 |  |  | NA (NA) — As pre-specified in protocol, Cmax was only calculated for participants with full PK samples. Thus, Cmax was not calculated for adolescent participants who only had sparse PK samples. | NA (NA) — As pre-specified in protocol, Cmax was only calculated for participants with full PK samples. Thus, Cmax was not calculated for adolescent participants who only had sparse PK samples.

13. Secondary Outcome: Observed Time to Reach Peak Plasma Concentration (Tmax) of Belumosudil
Description: Blood samples were collected at the specified timepoints to evaluate Tmax of belumosudil. As pre-specified in protocol, PK parameters were only calculated for participants with full PK samples. Thus, PK parameters were not calculated for adolescent participants who only had sparse PK samples.
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Median (Full Range); unit: Hours
Arm/Group | Adult Arm A: Belumosudil 200 mg QD | Adult Arm B: Belumosudil 200 mg BID | Adolescent Arm A: Belumosudil 200 mg QD | Adolescent Arm B: Belumosudil 200 mg BID
Number analyzed (Participants) | 5 | 5 | 2 | 1
Hours
  Cycle 1: number analyzed (Participants) | 5 | 5 | 0 | 0
  Cycle 1 | 2.90 [1.10 to 5.95] | 4.00 [1.18 to 7.75] |  |
  Cycle 2: number analyzed (Participants) | 4 | 4 | 2 | 1
  Cycle 2 | 1.98 [1.88 to 2.07] | 1.26 [1.00 to 4.03] | NA [NA to NA] — As pre-specified in protocol, Tmax was only calculated for participants with full PK samples. Thus, Tmax was not calculated for adolescent participants who only had sparse PK samples. | NA [NA to NA] — As pre-specified in protocol, Tmax was only calculated for participants with full PK samples. Thus, Tmax was not calculated for adolescent participants who only had sparse PK samples.
  Cycle 4: number analyzed (Participants) | 0 | 0 | 2 | 1
  Cycle 4 |  |  | NA [NA to NA] — As pre-specified in protocol, Tmax was only calculated for participants with full PK samples. Thus, Tmax was not calculated for adolescent participants who only had sparse PK samples. | NA [NA to NA] — As pre-specified in protocol, Tmax was only calculated for participants with full PK samples. Thus, Tmax was not calculated for adolescent participants who only had sparse PK samples.

14. Secondary Outcome: Area Under the Curve Over Time Interval From 0 to 6 Hours (AUC0-6) of Belumosudil
Description: Blood samples were collected at the specified timepoints to evaluate AUC0-6 of belumosudil. As pre-specified in protocol, PK parameters were only calculated for participants with full PK samples. Thus, PK parameters were not calculated for adolescent participants who only had sparse PK samples.
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*ng/mL
Arm/Group | Adult Arm A: Belumosudil 200 mg QD | Adult Arm B: Belumosudil 200 mg BID | Adolescent Arm A: Belumosudil 200 mg QD | Adolescent Arm B: Belumosudil 200 mg BID
Number analyzed (Participants) | 5 | 5 | 2 | 1
Hours*ng/mL
  Cycle 1: number analyzed (Participants) | 5 | 5 | 0 | 0
  Cycle 1 | 4430 (153) | 2380 (204) |  |
  Cycle 2: number analyzed (Participants) | 4 | 3 | 2 | 1
  Cycle 2 | 6860 (123) | 6520 (108) | NA (NA) — As pre-specified in protocol, AUC0-6 was only calculated for participants with full PK samples. Thus, AUC0-6 was not calculated for adolescent participants who only had sparse PK samples. | NA (NA) — As pre-specified in protocol, AUC0-6 was only calculated for participants with full PK samples. Thus, AUC0-6 was not calculated for adolescent participants who only had sparse PK samples.
  Cycle 4: number analyzed (Participants) | 0 | 0 | 2 | 1
  Cycle 4 |  |  | NA (NA) — As pre-specified in protocol, AUC0-6 was only calculated for participants with full PK samples. Thus, AUC0-6 was not calculated for adolescent participants who only had sparse PK samples. | NA (NA) — As pre-specified in protocol, AUC0-6 was only calculated for participants with full PK samples. Thus, AUC0-6 was not calculated for adolescent participants who only had sparse PK samples.

15. Secondary Outcome: Time to Response (TTR)
Description: TTR was measured as the time from first treatment to the time of first documentation of response.
Time Frame: From first dose of study drug to the time of first documentation of response or data cut-off, whichever occurred first(maximum duration: up to 40.5 months for adult arms and 27.6 months for adolescent arms)
Population: as for outcome 2
Measure: Median (Full Range); unit: Weeks
Arm/Group | Adult Arm A: Belumosudil 200 mg QD | Adult Arm B: Belumosudil 200 mg BID | Adolescent Arm A: Belumosudil 200 mg QD | Adolescent Arm B: Belumosudil 200 mg BID
Number analyzed (Participants) | 57 | 57 | 1 | 1
Weeks | 4.43 [3.7 to 80.1] | 4.43 [3.7 to 40.1] | 7.57 [7.5 to 7.6] | 4.14 [4.1 to 4.2]

16. Secondary Outcome: Time to Next Treatment (TTNT)
Description: The TTNT was measured as the time from first treatment to the time of new systemic cGVHD treatment, censored by last response assessment or long term follow up assessment, whichever was the latest and available.
Time Frame: From first dose of study drug to the time of new treatment or censoring date, whichever occurred first (maximum duration: up to 40.5 months for adult arms and 27.6 months for adolescent arms)
Population: mITT population included all randomized participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Adult Arm A: Belumosudil 200 mg QD | Adult Arm B: Belumosudil 200 mg BID | Adolescent Arm A: Belumosudil 200 mg QD | Adolescent Arm B: Belumosudil 200 mg BID
Number analyzed (Participants) | 77 | 75 | 2 | 1
Months | 24.2 [13.37 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of participants with events at study closure. | NA [14.55 to NA] — NA indicates that median and upper limit of CI was not estimable due to insufficient number of participants with events at study closure. | NA [NA to NA] — NA indicates that median and CI was not estimable due to insufficient number of participants with events at study closure. | 6.8 [NA to NA] — NA indicates that CI was not estimable due to insufficient number of participants with events at study closure.

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs): From first dose of study drug to the date of first documentation of progression or death due to any cause or data cut-off, whichever occurred first (maximum duration: up to 40.5 months for adult arms and 27.6 months for adolescent arms). All-cause mortality (deaths) were collected from first dose of study drug (Day 1) up to end of study, approximately 62 months.
Description: Safety population included all randomized participants who received at least one dose of study medication.
Groups:
- Adult Arm A: Belumosudil 200 mg QD: Participants received belumosudil 200 mg tablet orally QD in 28-day cycles until clinicallysignificant progression of cGVHD, histologic recurrence of underlying malignancy, unacceptabletoxicity, Investigator decision, participant preference/withdrawal of consent, loss of follow-up, sponsor decision, or death (whichever occurred first).
- Adult Arm B: Belumosudil 200 mg BID: Participants belumosudil 200 mg tablet orally BID in 28-day cycles until clinically significantprogression of cGVHD, histologic recurrence of underlying malignancy, unacceptable toxicity,Investigator decision, participant preference/withdrawal of consent, loss of follow-up, sponsor decision, or death (whichever occurred first).
- Adolescent Arm B: Belumosudil 200 mg BID: Participants received belumosudil 200 mg tablet orally BID in 28-day cycles until clinicallysignificant progression of cGVHD, histologic recurrence of underlying malignancy, unacceptabletoxicity, Investigator decision, participant preference/withdrawal of consent, loss of follow-up, sponsor decision, or death (whichever occurred first).
Arm/Group | Adult Arm A: Belumosudil 200 mg QD | Adult Arm B: Belumosudil 200 mg BID | Adolescent Arm A: Belumosudil 200 mg QD | Adolescent Arm B: Belumosudil 200 mg BID
All-Cause Mortality (participants affected / at risk) | 14/77 | 14/75 | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 36/77 | 30/75 | 1/2 | 0/1
Other Adverse Events (participants affected / at risk) | 73/77 | 73/75 | 2/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adult Arm A: Belumosudil 200 mg QD (N=77) | Adult Arm B: Belumosudil 200 mg BID (N=75) | Adolescent Arm A: Belumosudil 200 mg QD (N=2) | Adolescent Arm B: Belumosudil 200 mg BID (N=1)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cellulitis Orbital (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronavirus Infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Device Related Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large Intestine Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Listeriosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localised Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periorbital Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 7 (7) | 7 (8) | 1 (1) | 0 (0)
Rhinovirus Infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Septic Shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal Bacteraemia (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute Myeloid Leukaemia Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Microangiopathic Haemolytic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemic Hyperosmolar Nonketotic Syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Steroid Diabetes (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional State (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Mental Status Changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy Peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute Coronary Syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial Flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cardiac Failure Acute (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Enterovesical Fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumatosis Intestinalis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Face Oedema (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Multiple Organ Dysfunction Syndrome (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oedema Peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Liver Function Test Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Humerus Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Patella Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adult Arm A: Belumosudil 200 mg QD (N=77) | Adult Arm B: Belumosudil 200 mg BID (N=75) | Adolescent Arm A: Belumosudil 200 mg QD (N=2) | Adolescent Arm B: Belumosudil 200 mg BID (N=1)
Candida Infection (Infections and infestations) | 5 (7) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 6 (7) | 2 (2) | 0 (0) | 1 (1)
Coronavirus Infection (Infections and infestations) | 3 (3) | 6 (7) | 0 (0) | 0 (0)
Cytomegalovirus Infection Reactivation (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 5 (5) | 0 (0) | 0 (0)
Molluscum Contagiosum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis Externa (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 1 (4) | 1 (2)
Pneumonia (Infections and infestations) | 1 (1) | 6 (6) | 0 (0) | 0 (0)
Rhinovirus Infection (Infections and infestations) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
Skin Infection (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 17 (25) | 21 (25) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 7 (10) | 10 (18) | 0 (0) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Adrenal Insufficiency (Endocrine disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 13 (16) | 7 (10) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 7 (7) | 2 (2) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 13 (16) | 14 (26) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (4) | 7 (10) | 0 (0) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 (5) | 6 (7) | 1 (2) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (5) | 1 (1) | 1 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 4 (6) | 5 (8) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (6) | 7 (8) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (5) | 3 (5) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 6 (8) | 9 (10) | 0 (0) | 1 (1)
Confusional State (Psychiatric disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 4 (4) | 4 (4) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 6 (10) | 7 (7) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 7 (9) | 9 (10) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 4 (4) | 3 (4) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 22 (35) | 22 (30) | 1 (1) | 0 (0)
Neuropathy Peripheral (Nervous system disorders) | 5 (7) | 6 (8) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Peripheral Sensory Neuropathy (Nervous system disorders) | 4 (4) | 1 (2) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 2 (3) | 4 (7) | 0 (0) | 0 (0)
Dry Eye (Eye disorders) | 8 (9) | 5 (6) | 0 (0) | 0 (0)
Vision Blurred (Eye disorders) | 5 (5) | 4 (4) | 0 (0) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 4 (5) | 3 (3) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 3 (3) | 4 (5) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 4 (5) | 3 (3) | 0 (0) | 0 (0)
Hot Flush (Vascular disorders) | 2 (2) | 4 (5) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 13 (20) | 16 (32) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 22 (29) | 20 (29) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 25 (32) | 14 (18) | 1 (3) | 0 (0)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 4 (4) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (9) | 1 (1) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 11 (14) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 4 (5) | 1 (2) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 7 (9) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4) | 1 (2) | 0 (0)
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (6) | 0 (0) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 7 (11) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 13 (13) | 8 (13) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 8 (8) | 1 (2) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 8 (8) | 9 (10) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 33 (45) | 23 (40) | 0 (0) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 8 (8) | 9 (13) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 14 (19) | 4 (5) | 0 (0) | 1 (3)
Gastritis (Gastrointestinal disorders) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 7 (7) | 5 (5) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 24 (42) | 21 (25) | 1 (2) | 0 (0)
Oesophageal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 3 (4) | 4 (6) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 5 (6) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 22 (34) | 11 (12) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Dermatitis Psoriasiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (8) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (13) | 13 (14) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 7 (8) | 5 (6) | 0 (0) | 0 (0)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 3 (4) | 7 (10) | 0 (0) | 1 (1)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 7 (10) | 3 (3) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 (35) | 13 (19) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 9 (13) | 8 (9) | 0 (0) | 0 (0)
Knee Deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 12 (18) | 15 (17) | 2 (2) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 6 (10) | 4 (5) | 0 (0) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 3 (5) | 0 (0) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (5) | 0 (0) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 11 (12) | 14 (16) | 0 (0) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 4 (6) | 0 (0) | 0 (0) | 0 (0)
Chronic Kidney Disease (Renal and urinary disorders) | 1 (1) | 5 (6) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Premature Menopause (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Chills (General disorders) | 6 (8) | 3 (3) | 0 (0) | 0 (0)
Fatigue (General disorders) | 34 (49) | 23 (34) | 0 (0) | 0 (0)
Influenza Like Illness (General disorders) | 1 (1) | 6 (6) | 1 (1) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 4 (6) | 5 (5) | 0 (0) | 0 (0)
Oedema Peripheral (General disorders) | 22 (27) | 17 (22) | 0 (0) | 0 (0)
Pain (General disorders) | 4 (4) | 3 (5) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 14 (17) | 9 (10) | 1 (1) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 6 (14) | 12 (20) | 0 (0) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 7 (10) | 14 (28) | 1 (2) | 1 (1)
Blood Alkaline Phosphatase Increased (Investigations) | 5 (8) | 6 (12) | 0 (0) | 0 (0)
Blood Bicarbonate Decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood Cholesterol Increased (Investigations) | 3 (3) | 3 (3) | 1 (1) | 0 (0)
Blood Creatine Phosphokinase Increased (Investigations) | 3 (4) | 5 (5) | 0 (0) | 0 (0)
Blood Creatinine Increased (Investigations) | 6 (12) | 9 (20) | 0 (0) | 0 (0)
Blood Lactate Dehydrogenase Increased (Investigations) | 7 (8) | 8 (12) | 0 (0) | 1 (2)
Blood Urea Increased (Investigations) | 1 (2) | 4 (4) | 0 (0) | 0 (0)
Electrocardiogram Qt Prolonged (Investigations) | 2 (3) | 2 (2) | 1 (3) | 0 (0)
Gamma-Glutamyltransferase Increased (Investigations) | 7 (7) | 11 (20) | 0 (0) | 0 (0)
Lymphocyte Count Decreased (Investigations) | 2 (6) | 5 (8) | 0 (0) | 0 (0)
Platelet Count Decreased (Investigations) | 3 (4) | 5 (7) | 0 (0) | 0 (0)
Weight Decreased (Investigations) | 7 (16) | 8 (13) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 9 (10) | 6 (6) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 9 (11) | 13 (14) | 0 (0) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 4 (4) | 4 (4) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The sponsor decided to prematurely terminate the study due to the challenges encountered in recruiting adolescent participants. This decision was made without any safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2023-03-14): https://cdn.clinicaltrials.gov/large-docs/81/NCT03640481/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-26): https://cdn.clinicaltrials.gov/large-docs/81/NCT03640481/SAP_001.pdf